CLINICAL TRIAL: NCT02160743
Title: The Food Effect on Pharmacokinetics and Safety of Fixed-dose Combination of CJ-30056 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_ATM_104
Record Dates: First submitted 2014-05-28; First posted 2014-06-11 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Food Effect Study of CJ-30056 20mg/500mg
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ-30056 20mg/500mg (Experimental): fasting, fed
  Interventions: Dietary Supplement: CJ-30056 20/500mg (atorvastatin/metformin XR 20/500mg)
- group 2 (Experimental): fed, fasting
  Interventions: Dietary Supplement: CJ-30056 20/500mg (atorvastatin/metformin XR 20/500mg)

INTERVENTIONS:
Dietary Supplement: CJ-30056 20/500mg (atorvastatin/metformin XR 20/500mg)

SUMMARY:
This study evaluate the food effect on pharmacokinetics and safety of fixed-dose combination of "CJ-30056 20/500mg (atorvastatin/metformin XR 20/500mg)" in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Willing to adhere to protocol requirements and sign a informed consent form
2. Male volunteers in the age between 20 and 45 years old and have the weight range is not exceed ±20% of ideal weight
3. Subjects with no history of any significant chronic disease
4. Judged to be in good health on the basis of their vital sign, ECG, physical exam and routine laboratory data

Exclusion Criteria:

1. Use of barbital inducer or inhibitor medication within the 4 weeks before dosing
2. Symptom of an acute illness within 4 weeks prior to drug administration
3. History of clinically significant hepatic, renal, gastrointestinal diseases which might significantly interfere with ADME
4. History of surgery except or gastrointestinal diseases which might significantly change absorption of medicines
5. History of clinically significant allergies including drug allergies
6. History of clinically significant allergies about atorvastatin or metformin
7. Subjects who have ever or have plan to do intravenous injection of contrast medium (intravenous urography, intravenous cholangiography, computed tomography using contrast medium) within 28 days prior to drug administration
8. History of myopathy
9. Clinical laboratory test values are outside the accepted normal range

   * AST or ALT >1.25 times to normal range
   * Total bilirubin >1.5 times to normal range
   * e-GFR <90 mL/min
10. History of drug, caffein(caffein > 5 cups/day), smoking (cigarette > 10/day) or alcohol abuse(alcohol > 30 g/day)or Subjects who have ever drink within 7 days prior to drug administration
11. Special diet known to interfere with the absorption, distribution, metabolism or excretion of drugs (especially, consumption of grapefruit juice) within 7 days prior to drug administration
12. Donated blood within 60 days prior to dosing
13. Participated in a previous clinical trial within 60 days prior to dosing
14. Use of any other medication, including herbal products, within 10 days before dosing
15. Subjects considered as unsuitable based on medical judgement by investigators

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of atorvastatin | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36 hours post dose
Peak plasma concentration (Cmax) of metformin | 0, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24 hours post dose
area under the plasma concentration versus time curve (AUC0-t) of atorvastatin | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36 hours post dose
area under the plasma concentration versus time curve (AUC0-t) of metformin | 0, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24 hours post dose

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of 2-OH-atorvastatin | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36 hours post dose
Vz/F of atorvastatin and metformin | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36 hours post dose
area under the plasma concentration versus time curve (AUC0-t) of 2-OH-atorvastatin | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36 hours post dose
AUCinf of Atorvastatin, 2-OH-atorvastatin and metformin | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36 hours post dose
Tmax of Atorvastatin, 2-OH-atorvastatin and metformin | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36 hours post dose
t1/2β of Atorvastatin, 2-OH-atorvastatin and metformin | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36 hours post dose
CL/F of atorvastatin and metformin | 0, 0.33, 0.66, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 24, 36 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea